CLINICAL TRIAL: NCT00434330
Title: A Phase 2, Open-Label, Multi-Center, Dose Finding Study of the Safety, Pharmacodynamics, and Pharmacokinetics of Peginesatide for the Maintenance Treatment of Anemia in Hemodialysis Patients Previously Treated With Epoetin
Brief Title: Peginesatide for Maintenance Treatment of Anemia in Participants on Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-07; 2006-002815-28 (EudraCT Number)
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Anemia; Chronic Kidney Disease; Chronic Renal Failure
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemodialysis; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1, Q4W, SC, No Transition (Experimental)
  Interventions: Drug: peginesatide
- Cohort 2, Q4W, IV, No Transition (Experimental)
  Interventions: Drug: peginesatide
- Cohort 3, Q4W, SC, Transition (Experimental)
  Interventions: Drug: peginesatide
- Cohort 4, Q4W, IV, Transition (Experimental)
  Interventions: Drug: peginesatide
- Cohort 5, Q4W, SC, Transition (Experimental)
  Interventions: Drug: peginesatide
- Cohort 6, Q4W, IV, Transition (Experimental)
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: peginesatide — Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 milligram per kilogram (mg/kg) for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 7 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Cohort 1, Q4W, SC, No Transition
Drug: peginesatide — Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 mg/kg for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered intravenously (IV) once every 4 weeks for a total of 7 doses. No transition period between epoetin treatment and start of peginesatide treatment.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Cohort 2, Q4W, IV, No Transition
Drug: peginesatide — Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 mg/kg for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered subcutaneously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Cohort 3, Q4W, SC, Transition
Drug: peginesatide — Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 mg/kg for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered intravenously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Cohort 4, Q4W, IV, Transition
Drug: peginesatide — Tiered peginesatide starting doses of 0.04 mg/kg or 0.075 mg/kg for participants with an epoetin (alfa or beta) dose of ≤100 Units/kg/week or 100 to 150 Units/kg/week, respectively. Doses were administered subcutaneously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Cohort 5, Q4W, SC, Transition
Drug: peginesatide — Tiered peginesatide starting doses of 0.04 mg/kg or 0.075 mg/kg for participants with an epoetin (alfa or beta) dose of ≤100 Units/kg/week or 100 to 150 Units/kg/week, respectively. Doses were administered intravenously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Cohort 6, Q4W, IV, Transition

SUMMARY:
The purpose of this study was to determine the dose ranges of peginesatide administered intravenously or subcutaneously that maintained hemoglobin in participants on dialysis whose hemoglobin values were stable on epoetin (alfa or beta).

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents have been established as a treatment for anemia in subjects with chronic kidney disease, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia associated with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor, and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Six dose cohorts of 15 participants each were evaluated in this study. Participants received peginesatide injection once every 4 weeks administered intravenously or subcutaneously for a total of 7 doses.

ELIGIBILITY:
Inclusion Criteria:

* Participant is informed of the investigational nature of this study and has given written, witnessed informed consent in accordance with institutional, local, and national guidelines
* Males or females ≥ 18 years of age. Pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice a highly effective method of birth control for at least 4 weeks prior to study start, and must be willing to continue contraception until at least 4 weeks after the last dose of study drug
* Clinically stable on hemodialysis for ≥ 3 months prior to study start
* Epoetin (alfa or beta) maintenance therapy, ≥ 50 and ≤ 200 Units/kg/week, at the same dosing frequency, continuously prescribed for 8 weeks prior to study start
* Three mid- or end-of-week hemoglobin values of ≥ 10.0 and ≤ 12.5 grams per deciliter (g/dL) in the 4 weeks prior to study start, with ≤ 1.2 g/dL difference between any of the three values
* One transferrin saturation (TSAT) > 20% within 4 weeks prior to study start
* One ferritin level ≥ 100 ng/mL within 4 weeks prior to study start
* One serum or red cell folate level ≥ lower limit of normal during the 4 weeks prior to study start
* One vitamin B12 level ≥ lower limit of normal during the 4 weeks prior to study start
* One C-reactive protein (CRP) level ≤ 30 mg/L within 4 weeks prior to study start
* Urea clearance/volume (Kt/V) ≥ 1.2 within 4 weeks prior to study start
* One white blood cell count (WBC) ≥ 3.0 x 10^9/L within 4 weeks prior to study start
* One platelet count ≥ 100 x 10^9/L and ≤ 500 x 10^9/L within 4 weeks prior to study start

Exclusion Criteria:

* Pregnant or breast-feeding participants
* Known intolerance to any erythropoiesis stimulating agent, parenteral iron supplementation or pegylated molecules
* History of antibodies to any erythropoiesis stimulating agent or history of pure red cell aplasia (PRCA)
* Known bleeding or coagulation disorder
* Known hematologic disease (e.g., homozygous sickle-cell disease, thalassemia of all types, multiple myeloma, hemolytic anemia)
* Uncontrolled or symptomatic inflammatory disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, etc.)
* Known history of seizure disorder or received anti-epileptic medication within the previous 6 months
* Uncontrolled or symptomatic secondary hyperparathyroidism, per Investigator's clinical judgment
* Poorly controlled hypertension within 4 weeks prior to study start, per Investigator's clinical judgment
* Chronic congestive heart failure of New York Heart Association class III or IV
* High likelihood of early withdrawal or interruption of the study (e.g., myocardial infarction, severe or unstable coronary artery disease, stroke, respiratory, autoimmune, neuropsychiatric, or neurological abnormalities, liver disease including active hepatitis B or C, active HIV disease, or any other clinically significant medical diseases or conditions in the prior 6 months that may, in the Investigator's opinion, interfere with safety, assessment, or follow-up of the participant)
* Evidence of malignancy within the past 5 years (except non-melanoma skin cancer which is not an exclusion criterion)
* Life expectancy < 12 months
* Temporary (untunneled) dialysis access catheter
* Anticipated elective surgery during the study period, that may be expected to lead to significant blood loss, including vascular access surgery such as an arteriovenous fistula or graft, or a scheduled kidney transplant
* Red blood cell or whole blood transfusion within 12 weeks prior to study start
* Received antibiotics for systemic infection within 2 weeks prior to study start
* Previous exposure to any investigational agent within 6 weeks prior to study start, or planned receipt of an investigational agent, other than as specified by this protocol, during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2006-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax, Inc.
Locations (13):
- Bulgaria (7):
  - Research Facility, Burgas
  - Research Facility, Pleven
  - Research Facility, Plovdiv
  - Research Facility, Rousse
  - Research Facility, Sofia
  - Research Facility, Varna
  - Research Facility, Veliko Tarnovo
- Romania (5):
  - Research Facility, Arad
  - Research Facility, Bacau
  - Research Facility, Bucharest
  - Research Facility, Iași
  - Research Facility, Timișoara
- Research Facility, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Q4W, SC, No Transition: Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 milligram per kilogram (mg/kg) for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 7 doses. No transition period between epoetin treatment and start of peginesatide treatment.
- Cohort 2, Q4W, IV, No Transition: Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 mg/kg for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered intravenously (IV) once every 4 weeks for a total of 7 doses. No transition period between epoetin treatment and start of peginesatide treatment.
- Cohort 3, Q4W, SC, Transition: Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 mg/kg for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered subcutaneously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
- Cohort 4, Q4W, IV, Transition: Tiered peginesatide starting doses of 0.05, 0.075, or 0.1 mg/kg for participants on an epoetin (alfa or beta) dose of ≤100 Units/kg/week, >100 to 150 Units/kg/week, or >150 Units/kg/week, respectively. Doses were administered intravenously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
- Cohort 5, Q4W, SC, Transition: Tiered peginesatide starting doses of 0.04 mg/kg or 0.075 mg/kg for participants with an epoetin (alfa or beta) dose of ≤100 Units/kg/week or 100 to 150 Units/kg/week, respectively. Doses were administered subcutaneously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
- Cohort 6, Q4W, IV, Transition: Tiered peginesatide starting doses of 0.04 mg/kg or 0.075 mg/kg for participants with an epoetin (alfa or beta) dose of ≤100 Units/kg/week or 100 to 150 Units/kg/week, respectively. Doses were administered intravenously once every 4 weeks for a total of 7 doses. With transition period between epoetin treatment and start of peginesatide treatment.
Period: Overall Study
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition
Started | 15 | 15 | 16 | 15 | 15 | 15
Completed | 14 | 15 | 13 | 13 | 14 | 14
Not Completed | 1 | 0 | 3 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Renal transplant | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Not Compliant With Study | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition | Total
Number analyzed (Participants) | 15 | 15 | 16 | 15 | 15 | 15 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 12 | 13 | 12 | 12 | 70
  >=65 years | 4 | 5 | 4 | 2 | 3 | 3 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.42) | 58.1 (13.91) | 46.1 (17.22) | 50.4 (12.47) | 51.1 (11.43) | 53 (13.22) | 51.9 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 5 | 4 | 6 | 4 | 34
  Male | 6 | 9 | 11 | 11 | 9 | 11 | 57

OUTCOME MEASURES:

1. Primary Outcome: Mean Hemoglobin Throughout the Trial and Mean Hemoglobin Change From Baseline Throughout the Trial.
Description: The Baseline hemoglobin was the mean of the four most recent mid- or end-of-week predialysis hemoglobin values collected prior to study start. Study start was the date of the first dose of peginesatide injection in participants who did not have a one-week transition period, or the date when Epoetin treatment was first withheld in participants who did have a one-week transition period.
Time Frame: Baseline and Weeks 2-29
Population: Modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
g/dL
  Baseline [N=15, 15, 14, 15, 15, 15] | 11.10 (0.600) | 11.34 (0.596) | 11.42 (0.448) | 11.19 (0.628) | 11.11 (0.810) | 11.24 (0.742)
  Weeks 2-29 [N=15, 15, 15, 15, 15, 15] | 11.64 (0.722) | 11.57 (0.771) | 11.98 (0.858) | 11.86 (0.538) | 11.92 (0.699) | 11.19 (1.114)
  Change from Baseline [N=15, 15, 14, 15, 15, 15] | 0.53 (0.600) | 0.23 (0.776) | 0.57 (0.793) | 0.67 (0.752) | 0.82 (0.935) | -0.05 (1.000)

2. Other Pre Specified Outcome: Proportion of Participants With Hemoglobin Within 1.0 g/dL Below Baseline to 1.5 g/dL Above Baseline Throughout the Trial (Weeks 2-29)
Description: Hemoglobin relative to baseline: Hemoglobin at a given time point was considered to be not within the specified range (within 1 g/dL below to 1.5 g/dL above baseline) if the hemoglobin value at the time point was not within the range and the next available hemoglobin value within 14 days after the time point also was not within the specified range. These calculations were determined for all time points within a specified time period.
Time Frame: Weeks 2 to 29
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
percentage of participants | 0.267 | 0.133 | 0.200 | 0.333 | 0.400 | 0.267

3. Other Pre Specified Outcome: Proportion of Participants Who Maintained Hemoglobin Within 10 to 12.5 g/dL Throughout the Trial
Description: Hemoglobin relative to baseline: Hemoglobin at a given time point was considered to be not within the specified range (within the range of 10 g/dL to 12.5 g/dL) if the hemoglobin value at the time point was not within the range and the next available hemoglobin value within 14 days after the time point also was not within the specified range. These calculations were determined for all time points within a specified time period.
Time Frame: Weeks 2 to 29
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
percentage of participants | 0.333 | 0.200 | 0.200 | 0.200 | 0.200 | 0.067

4. Other Pre Specified Outcome: Proportion of Participants Who Maintain Hemoglobin Within 9.5 to 13.0 g/dL Throughout the Trial
Description: Hemoglobin relative to baseline: Hemoglobin at a given time point was considered to be not within the specified range (within the range of 9.5 g/dL to 13.0 g/dL) if the hemoglobin value at the time point was not within the range and the next available hemoglobin value within 14 days after the time point also was not within the specified range. These calculations were determined for all time points within a specified time period.
Time Frame: Weeks 2 to 29
Population: mITT population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
percentage of participants | 0.800 | 0.667 | 0.533 | 0.533 | 0.600 | 0.600

ADVERSE EVENTS:
Arm/Group | Cohort 1, Q4W, SC, No Transition | Cohort 2, Q4W, IV, No Transition | Cohort 3, Q4W, SC, Transition | Cohort 4, Q4W, IV, Transition | Cohort 5, Q4W, SC, Transition | Cohort 6, Q4W, IV, Transition
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/15 | 3/16 | 1/15 | 3/15 | 2/15
Other Adverse Events (participants affected / at risk) | 10/15 | 8/15 | 7/16 | 8/15 | 10/15 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Q4W, SC, No Transition (N=15) | Cohort 2, Q4W, IV, No Transition (N=15) | Cohort 3, Q4W, SC, Transition (N=16) | Cohort 4, Q4W, IV, Transition (N=15) | Cohort 5, Q4W, SC, Transition (N=15) | Cohort 6, Q4W, IV, Transition (N=15)
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Penile necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Q4W, SC, No Transition (N=15) | Cohort 2, Q4W, IV, No Transition (N=15) | Cohort 3, Q4W, SC, Transition (N=16) | Cohort 4, Q4W, IV, Transition (N=15) | Cohort 5, Q4W, SC, Transition (N=15) | Cohort 6, Q4W, IV, Transition (N=15)
Vertigo (Ear and labyrinth disorders) | 4 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 2 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 3 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 4 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 1
Chest pain (General disorders) | 0 | 3 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 3 | 1 | 0 | 2 | 1
Tracheobronchitis (Infections and infestations) | 3 | 1 | 0 | 0 | 2 | 1
Tooth abscess (Infections and infestations) | 2 | 0 | 0 | 1 | 2 | 0
Hepatitis C (Infections and infestations) | 0 | 3 | 0 | 2 | 0 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 3 | 3 | 3 | 1 | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 1 | 1 | 1
Procedural headache (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 3 | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 3 | 4 | 3
Blood pressure increased (Investigations) | 4 | 0 | 2 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2 | 4 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 9 | 4 | 7 | 4 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 2 | 0
Hypotension (Vascular disorders) | 6 | 5 | 2 | 2 | 2 | 2
Hypertensive crisis (Vascular disorders) | 4 | 6 | 2 | 5 | 0 | 4
Hypertension (Vascular disorders) | 2 | 2 | 4 | 4 | 1 | 0

LIMITATIONS AND CAVEATS:
Notable issues with some documentation occurred at some of the study sites. In general, overall results excluding the sites with issues were comparable to results based on the full population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications may not contain Sponsor confidential information, and will be subject to Sponsor review prior to submission for publication.